CLINICAL TRIAL: NCT03412136
Title: Acute Decrease in Serum Testosterone After Glucose and Protein Beverages in Adolescent Males
Brief Title: The Acute Effect of Protein or Carbohydrate Intake on Testosterone Levels and Food Intake in Children and Adolescent Boys
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, G. Harvey Anderson, Full Professor, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 29191
Record Dates: First submitted 2018-01-06; First posted 2018-01-26 (Actual); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Appetitive Behavior; Pediatric Obesity
Keywords: Testosterone; Food Intake; Appetite
MeSH Terms: conditions — Appetitive Behavior; Pediatric Obesity | interventions — Glucose; Proteins

STUDY DESIGN:
Intervention Model Description: In a randomized, crossover study, sixteen 9-18 y old males were given beverages containing either: 1) whey protein (1g/kg bodyweight), 2) glucose (1g/kg bodyweight) or a calorie-free control (C). Serum testosterone, appetite biomarkers and subjective appetite were measured prior (0) and at 20, 35 and 65 minutes after the consumption of the beverage. Food intake at an ad libitum pizza meal was assessed 20 min later (65-85min).
Who Masked: Participant
Masking Description: The experimental beverages contained either 1g of glucose monohydrate (BioShop Canada Inc., Burlington, Ontario, Canada) or 1g of protein (plain whey-protein isolate; BiPro USA., Eden Prairie, Minnesota, U.S.A) per kg of bodyweight. A non-calorie drink was used as control. All beverages were flavoured with 1.5ml of chocolate extract (Vanilla Food Company, Markham, Ontario, Canada) to account for the flavor differences and mixed with 500ml of water. The whey protein and control beverages were sweetened with 0.2g sucralose (Tate & Lyle, Stoney Creek, Ontario, Canada) in order to match sweetness with the glucose beverage.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Experimental)
  Interventions: Dietary Supplement: Control
- Glucose (Experimental)
  Interventions: Dietary Supplement: Glucose
- Protein (Experimental)
  Interventions: Dietary Supplement: Protein

INTERVENTIONS:
Dietary Supplement: Control — Participants were given 5 minutes to ingest the non-caloric beverage which contained 1.5ml of chocolate extract (Vanilla Food Company, Markham, Ontario, Canada) to account for the flavor differences and mixed with 500ml of water and sweetened with 0.2g sucralose (Tate & Lyle, Stoney Creek, Ontario, Canada) in order to match sweetness with the glucose beverage.
  Arms: Control
Dietary Supplement: Glucose — Participants were given 5 minutes to ingest the beverage which contained either 1g of protein (plain whey-protein isolate; BiPro USA., Eden Prairie, Minnesota, U.S.A) per kg of bodyweight and was flavoured with 1.5ml of chocolate extract (Vanilla Food Company, Markham, Ontario, Canada) to account for the flavor differences and mixed with 500ml of water.
  Arms: Glucose
Dietary Supplement: Protein — Participants were given 5 minutes to ingest the beverage which contained 1g of glucose monohydrate (BioShop Canada Inc., Burlington, Ontario, Canada) per kg of bodyweight and flavoured with 1.5ml of chocolate extract (Vanilla Food Company, Markham, Ontario, Canada) to account for the flavor differences and mixed with 500ml of water.
  Arms: Protein

SUMMARY:
The purpose of this study was to determine the effect of acute protein and glucose intake on testosterone levels measured in adolescent boys and determine whether changes in testosterone levels are associated with alterations in short-term food intake. It was hypothesized that 1) ingestion of a protein beverage would result in no change of testosterone levels whereas glucose would result in a significant decrease of testosterone levels 60 minutes after ingestion and 2) decreases of testosterone levels as a result of the glucose preload would predict food intake for boys of similar body size. The first objective was to investigate the effect of an acute protein or glucose drink on testosterone levels and the second objective was to determine whether changes of testosterone levels associate with food intake.

ELIGIBILITY:
Inclusion Criteria:

* 9-18 years, healthy, male.

Exclusion Criteria:

* History of prematurity, chronic illness, were taking any medications known to affect glucose homeostasis, appetite or pubertal development.

Ages: 9 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Normal weight and overweight/obese adolescent males (n=34) age 9 to 18 were recruited via print advertisement in the local Toronto newspaper. verweight was categorized as in the 85th-95th percentile and obesity in ≥95th percentile.
Enrollment: 34 (Actual)
Dates: Start 2014-03-08 (Actual); Primary Completion 2016-04-10 (Actual); Study Completion 2016-04-10 (Actual)

PRIMARY OUTCOMES:
Testosterone Change | 0-65 minutes
  The first blood draw was taken prior to ingesting the experimental beverage at baseline (0 minutes). Participants were then given 5 minutes to ingest the beverage, and blood was later obtained 20, 35 and 65 minutes after baseline blood draw. Units were measured in ng/dl.

SECONDARY OUTCOMES:
Appetite Biomarkers- Glucose | 0-85 minutes
  Glucose. Units were measured in mg/dl.
Appetite Biomarkers- Glucagon-like peptide-1 | 0-85 minutes
  Glucagon-like peptide-1. Units were measured in pM.
Appetite Biomarkers- Active Ghrelin | 0-85 minutes
  Active Ghrelin. Units were measured in pg/ml.
Appetite Biomarkers- Insulin | 0-85 minutes
  Insulin. Units were measured in uIu/ml.
Subjective Appetite- Determination to eat | 0-85 minutes
  Visual Analog Scales were employed to assess subjective appetite based on the Determination to Eat. Units were measured in mm (based on a 100mm scale).
Subjective Appetite- Hunger | 0-85 minutes
  Visual Analog Scales were employed to assess subjective appetite based on feelings of Hunger. Units were measured in mm (based on a 100mm scale).
Subjective Appetite- Fullness | 0-85 minutes
  Visual Analog Scales were employed to assess subjective appetite based on feelings of FullnessUnits were measured in mm (based on a 100mm scale).
Subjective Appetite- Prospective Food Consumption | 0-85 minutes
  Visual Analog Scales were employed to assess subjective appetite based on Prospective Food Consumption. Units were measured in mm (based on a 100mm scale).
Food Intake | 65-85 minutes
  Participants were provided an ad libitum pizza meal. The participants were instructed to eat during the next 20 min until they were comfortably full. Based on the participant preferences determined during screening, two varieties of Deep 'N Delicious 5-inch-diameter pizza were provided for consumption; pepperoni and three-cheese pizzas (McCain Canada Ltd., Florenceville, Ontario, Canada). Units were measuring in kcal.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available to other researchers.Participant's identities will be kept confidential. Records will be kept in a locked filing cabinet in the Fitzgerald building at 150 College Street, room 305. Access will be restricted to those directly involved with the project, such as the investigator and the co-investigators. Following recruitment and attainment of informed consent, participants will be given an ID # which will be used on all forms and data analysis. Informed consent forms will be kept in a locked cabinet in a locked office, contain participant names. Research records will be identified by initials, ID number, test and date. Results identified by date and ID number will only be entered on password-protected personal computers kept in locked laboratories or offices at the University of Toronto. Any electronic data will be held on encrypted computers and USB sticks for the same period of time.

REFERENCES:
- [Background] Schwartz A, Patel BP, Vien S, McCrindle BW, Anderson GH, Hamilton J. Acute decrease in serum testosterone after a mixed glucose and protein beverage in obese peripubertal boys. Clin Endocrinol (Oxf). 2015 Sep;83(3):332-8. doi: 10.1111/cen.12630. Epub 2014 Nov 27. PMID 25308907
- [Background] Anderson KE, Rosner W, Khan MS, New MI, Pang SY, Wissel PS, Kappas A. Diet-hormone interactions: protein/carbohydrate ratio alters reciprocally the plasma levels of testosterone and cortisol and their respective binding globulins in man. Life Sci. 1987 May 4;40(18):1761-8. doi: 10.1016/0024-3205(87)90086-5. PMID 3573976
- [Background] Caronia LM, Dwyer AA, Hayden D, Amati F, Pitteloud N, Hayes FJ. Abrupt decrease in serum testosterone levels after an oral glucose load in men: implications for screening for hypogonadism. Clin Endocrinol (Oxf). 2013 Feb;78(2):291-6. doi: 10.1111/j.1365-2265.2012.04486.x. PMID 22804876
- [Background] Anderson GH, Hunschede S, Akilen R, Kubant R. Physiology of Food Intake Control in Children. Adv Nutr. 2016 Jan 15;7(1):232S-240S. doi: 10.3945/an.115.009357. Print 2016 Jan. PMID 26773031
- [Result] Konforte D, Shea JL, Kyriakopoulou L, Colantonio D, Cohen AH, Shaw J, Bailey D, Chan MK, Armbruster D, Adeli K. Complex biological pattern of fertility hormones in children and adolescents: a study of healthy children from the CALIPER cohort and establishment of pediatric reference intervals. Clin Chem. 2013 Aug;59(8):1215-27. doi: 10.1373/clinchem.2013.204123. Epub 2013 May 1. PMID 23637248
- [Result] Du M, Shen QW, Zhu MJ, Ford SP. Leucine stimulates mammalian target of rapamycin signaling in C2C12 myoblasts in part through inhibition of adenosine monophosphate-activated protein kinase. J Anim Sci. 2007 Apr;85(4):919-27. doi: 10.2527/jas.2006-342. Epub 2006 Dec 18. PMID 17178807
- [Result] Caufriez A. The pubertal spurt: effects of sex steroids on growth hormone and insulin-like growth factor I. Eur J Obstet Gynecol Reprod Biol. 1997 Feb;71(2):215-7. doi: 10.1016/s0301-2115(96)02638-3. PMID 9138969
- [Derived] Schwartz A, Hunschede S, Lacombe RJS, Chatterjee D, Sanchez-Hernandez D, Kubant R, Bazinet RP, Hamilton JK, Anderson GH. Acute decrease in plasma testosterone and appetite after either glucose or protein beverages in adolescent males. Clin Endocrinol (Oxf). 2019 Aug;91(2):295-303. doi: 10.1111/cen.14005. Epub 2019 May 16. PMID 31055857